CLINICAL TRIAL: NCT00003219
Title: A Phase II Trial of Perillyl Alcohol (NSC 641066) Administered Daily in Patients With Metastatic Breast Cancer
Brief Title: Perillyl Alcohol in Treating Patients With Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000066080; R21CA072500 (NIH); WCCC-CO-9611; NCI-T97-0068
Record Dates: First submitted 1999-11-01; First posted 2004-07-19 (Estimated); Last update posted 2019-12-13 (Actual); Status verified 2012-10

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — perillyl alcohol

INTERVENTIONS:
Drug: perillyl alcohol

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of perillyl alcohol in treating patients with metastatic breast cancer that has not responded to previous chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the clinical effectiveness (i.e., objective tumor response, time to treatment failure, and survival) of perillyl alcohol in patients with previously treated metastatic breast cancer. II. Define the acute and chronic toxic effects of perillyl alcohol in this patient population.

OUTLINE: Patients are given oral perillyl alcohol 4 times per day. Dose escalation of perillyl alcohol may occur in individual patients if no unacceptable toxicity is observed. Treatment is continued as long as the patient benefits from treatment, does not show progressive disease, and does not experience irreversible or life threatening toxicity. Patients are evaluated for response monthly while receiving treatment on this study. Patients are followed at 2-4 weeks after the last treatment.

PROJECTED ACCRUAL: Approximately 40 patients will be accrued over 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Microscopically confirmed metastatic breast cancer Must be refractory or have recurred after at least 1 systemic chemotherapy regimen Estrogen receptor positive tumors must have failed or recurred after hormonal therapy At least 1 site of measurable disease required Previously radiated lesions are not considered measurable unless there is evidence of disease progression after completion of radiation therapy No known brain metastases Hormone receptor status: Unspecified

PATIENT CHARACTERISTICS: Age: 18 and over Menopausal status: Not specified Performance status: Zubrod 0-2 Life expectancy: At least 12 weeks Hematopoietic: WBC at least 4000/mm3 Platelet count at least 100,000/mm3 Absolute neutrophil count at least 1500/mm3 Hepatic: Bilirubin no greater than 1.5 mg/dL SGOT no greater than 2 times normal Renal: Creatinine no greater than 1.5 mg/dL BUN no greater than 30 mg/dL Other: Effective birth control must be used by fertile patients (barrier method preferred) Not pregnant or nursing

PRIOR CONCURRENT THERAPY: Recovered from toxic effects of prior treatment Biologic therapy: No immunologic therapy within the past 2 weeks Chemotherapy: No chemotherapy within the past 4 weeks (6 weeks for mitomycin or nitrosoureas) See Disease Characteristics Endocrine therapy: No hormonal therapy within the past 2 weeks See Disease Characteristics Radiotherapy: No radiotherapy within the past 4 weeks See Disease Characteristics Surgery: Not specified Other: No concurrent cholesterol lowering agents, supplemental vitamins, or other antioxidants

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-05; Primary Completion 1998-05 (Actual); Study Completion 1998-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard H. Bailey, MD, Study Chair — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin, United States

REFERENCES:
- [Result] Bailey HH, Attia S, Love RR, Fass T, Chappell R, Tutsch K, Harris L, Jumonville A, Hansen R, Shapiro GR, Stewart JA. Phase II trial of daily oral perillyl alcohol (NSC 641066) in treatment-refractory metastatic breast cancer. Cancer Chemother Pharmacol. 2008 Jun;62(1):149-57. doi: 10.1007/s00280-007-0585-6. Epub 2007 Sep 21. PMID 17885756